CLINICAL TRIAL: NCT01261416
Title: Pharmacokinetics and Safety of IV Levetiracetam (Keppra) in Full Term and Preterm Neonates
Brief Title: Pharmacokinetics of Levetiracetam (Keppra) in Neonates
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Stephanie Merhar MD, Cincinnati Children's Hospital Medical Center
Other Study IDs: 101335-2
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Seizures; Epilepsy
Keywords: seizures; epilepsy; neonatal; levetiracetam
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants with seizures
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — Patients will receive levetiracetam as needed for clinical and/or electrographic seizures. Need for levetiracetam will be determined by the clinical team and will NOT determined by the study protocol.

SUMMARY:
The primary objective of this study is to determine the pharmacokinetic profile of a loading dose of intravenous levetiracetam, given for clinical reasons, in term and late preterm infants with seizures. Secondary objectives are to evaluate the safety and efficacy of levetiracetam in term and preterm infants with seizures.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 32 weeks
* Postnatal age ≤ 30 days
* Birth weight ≥ 2000 grams
* Admitted to the NICU at Cincinnati Children's Hospital or Good Samaritan Hospital
* Clinical or electrographic seizures of any etiology
* Seizures or seizure prophylaxis requiring treatment with levetiracetam
* Parental consent obtained

Exclusion Criteria:

* Infants with renal insufficiency indicated by serum creatinine > 2.0 at any time
* Infants who have previously received levetiracetam
* Parents refuse consent
* Attending physician does not wish the infant to be enrolled in the study
* Infants who are currently receiving an investigational drug

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants ≥ 32 weeks gestation and ≤ 30 days of age requiring treatment with levetiracetam for clinical and/or electrographic seizures or seizure prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | 24 hours after dose
  Blood specimens for quantitation of levetiracetam and its metabolite L057 will be obtained from an indwelling vascular catheter not used for study drug infusion or by heel stick in three different sampling schedules:
  Group 1 (n=6): at times 2-15 minutes after the end of infusion, 1-2 hours, and 12 hours post start of infusion Group 2 (n=6): at times 2-15 minutes after the end of infusion, 2-4 hours, and 18 hours post start of infusion Group 3 (n=6): at times 2-15 minutes after the end of infusion, 4-8 hours, and 20-24 hours post start of infusion

SECONDARY OUTCOMES:
Change in vital sign baseline | 24 hours
  Short term treatment-emergent adverse effects of levetiracetam will be measured by change from vital sign baseline in the 24 hours after the dose.
Number of participants with adverse events | 24 hours
  Participants' medical records will be reviewed for any adverse effects of the medication seen in the 24 hours after the loading dose.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Merhar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States